CLINICAL TRIAL: NCT03750591
Title: Observational Study on Effectiveness and Safety of Integrative Korean Medicine Treatment for Inpatients With Sciatica Due to Lumbar Intervertebral Disc Herniation
Status: Completed | Type: Observational
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Principal Investigator, In-Hyuk Ha, KMD, Director, Jaseng Medical Foundation
Other Study IDs: JS-CT-2017-05-1
Record Dates: First submitted 2018-11-14; First posted 2018-11-23 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Sciatica Due to Intervertebral Disc Disorder; Intervertebral Disc Displacement; Sciatica; Sciatic Radiculopathy
Keywords: Integrative Korean medicine; treatment; effectiveness; safety; Lumbar intervertebral disc herniation
MeSH Terms: conditions — Intervertebral Disc Displacement; Sciatica | interventions — Phytotherapy; Acupuncture Therapy; Electroacupuncture; Cupping Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Integrative Korean medicine treatment group: Observation of pain, function, quality of life, satisfaction, and adverse events in inpatients with lumbar intervertebral disc herniation hospitalized at 4 Korean medicine hospitals
  Interventions:
  Drug: Herbal medicine Procedure/Surgery: Chuna manual therapy Procedure/Surgery: Bee venom pharmacopuncture Procedure/Surgery: Pharmacopuncture Procedure/Surgery: Acupuncture Procedure/Surgery: Electroacupuncture Procedure/Surgery: Cupping Other intervention(s)
  Interventions: Drug: Herbal medicine; Procedure: Chuna manual therapy; Procedure: Bee venom pharmacopuncture; Procedure: Pharmacopuncture; Procedure: Acupuncture; Procedure: Electroacupuncture; Procedure: Cupping; Other: Other intervention(s)

INTERVENTIONS:
Drug: Herbal medicine — Herbal medicine will be mainly administered in water-based decoction (120ml) and dried powder (2g) form (the ingredients are mainly, but not restricted to: Ostericum koreanum, Eucommia ulmoides, Acanthopanax sessiliflorus, Achyranthes japonica, Psoralea corylifolia, Saposhnikovia divaricata, Cibotium barometz, Lycium chinense, Boschniakia rossica, Cuscuta chinensis, Glycine max, Atractylodes japonica).
  Other Names: Traditional herbal medicine
Procedure: Chuna manual therapy — Chuna is a Korean spinal manipulation that incorporates spinal manipulation techniques for joint mobilization involving highvelocity, low amplitude thrusts to joints slightly beyond the passive range of motion and gentle force to joints within the passive range of movement.
  Chuna manipulation will be administered at the physician's discretion.
  Other Names: Chuna manipulation; Chuna spinal manipulation
Procedure: Bee venom pharmacopuncture — Bee venom pharmacopuncture will be administered only after confirming a negative response to hypersensitivity skin test.
  Diluted bee venom (saline:bee venom ratio, 10,000:1) filtered for allergens will be injected at 4-5 acupoints proximal to the dysfunctional site at the physician's discretion. Each acupuncture point will be injected to a total of 0.5-1 cc using disposable injection needles (CPL, 1 cc, 26gauze(G) x 1.5 syringe, Shinchang medical co., Korea).
  Other Names: Bee venom acupuncture
Procedure: Pharmacopuncture — Pharmacopuncture consisting of select herbal ingredients will be administered at Ah-shi points and local acupuncture points using disposable injection needles (CPL, 1 cc, 26gauze(G) x 1.5 syringe, Shinchang medical co., Korea).
Procedure: Acupuncture — Acupuncture treatment will be administered using mainly proximal acupuncture points and Ah-shi points.
Procedure: Electroacupuncture — Electroacupuncture treatment will be administered using mainly proximal acupuncture points and Ah-shi points.
Procedure: Cupping — Cupping treatment will be administered at 1-2 points using mainly proximal acupuncture points and Ah-shi points.
Other: Other intervention(s) — Patients will be allowed any other additional intervention(s) as deemed necessary by the attending physician regardless of type or dose, and patterns of use will be investigated and recorded as an pragmatic clinical study.

SUMMARY:
Observational study on the effectiveness and safety of integrative Korean medicine treatment for inpatients with sciatica due to lumbar intervertebral disc herniation

DETAILED DESCRIPTION:
Establishment of a Korean medicine inpatient treatment registry of inpatients with sciatica due to lumbar intervertebral disc herniation with or without spinal stenosis, in conjunction with an observational study to the aim of evaluating the effectiveness and safety of Korean medicine treatment for inpatients

ELIGIBILITY:
Inclusion Criteria:

1. Lumbar intervertebral disc herniation as confirmed by a doctor of medicine or a doctor of Korean medicine through an MRI taken within 3 years
2. Patients with radiculopathy (ipsilateral or bilateral radiculopathy)
3. Patients whose pain intensity of back pain or radiating leg pain is NRS≥5
4. Patients aged 19 to 70
5. Patients who have agreed to participate in the clinical study and given written informed consent
6. Patients admitted to a Korean medicine hospital for treatment

Exclusion Criteria:

1. Patients who have been diagnosed with a serious disease that may cause low back pain or neck pain (e.g. spinal metastasis of tumor, acute fracture, spinal dislocation)
2. Patients admitted due to pain caused by traffic accidents
3. Patients with progressive neurological deficit or severe neurological symptoms such as spinal cord injury
4. Patients with severe mental illness
5. Patients with difficulty or refusal to give sign written informed consent
6. Patients for whom the researchers judge participation in the clinical study to be difficult
7. Diagnosis of lumbar spondylolisthesis of Meyerding Ⅱ or higher by a doctor of medicine or doctor of Korean medicine through X-ray or MRI

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are admitted or scheduled to be admitted to Jaseng Hospital of Korean Medicine, Bucheon Jaseng Hospital of Korean Medicine, Daejeon Jaseng Hospital of Korean Medicine, or Haeundae Jaseng Hospital of Korean Medicine
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2018-03-31 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2019-11-08 (Actual)

PRIMARY OUTCOMES:
NRS change from Baseline NRS at discharge | Baseline (admission), discharge (up to 14 weeks after baseline)
  Numeric rating scale (NRS) of low back pain, and radiating leg pain In pain measurement using NRS, patients are asked to rate their pain by selecting a number from 0 to 10 that best represents their pain severity between the anchors of 0 which indicates 'no pain', and 10 which indicates 'worst pain possible'.
ODI change from Baseline ODI at discharge | Baseline (admission), discharge (up to 14 weeks after baseline)
  Oswestry Disability Index(ODI) The ODI evaluates functional impairment and is a 10-item questionnaire developed to assess the level of disability due to back pain. Each item is graded into 6 levels, each representing a score of 0-5. Higher scores indicate greater limitation relating to back pain.
PGIC | 6 months after baseline
  Patient global impression of change (PGIC) PGIC grades the level of subjective improvement into 7 levels (1, very much improved; 2, much improved; 3, slightly improved; 4, no change; 5, slightly worse; 6, much worse; and 7, very much worse).

SECONDARY OUTCOMES:
EQ-5D change from Baseline EQ-5D at each time point | Baseline (admission), 2 weeks after baseline, discharge (up to 14 weeks after baseline), 6 months after baseline
  EuroQol-5 Dimension(EQ-5D) EQ-5D is a tool developed for health-related quality of life (HRQoL) assessment, and is widely used in the health care sector. Scores range from -1, 'health worse than death' to 1, 'perfect health'. EQ-5D-5L has 5 dimensions covering current health status and functionality: mobility (M), self care (SC), usual activities (UA), pain/discomfort (PD), and anxiety/depression (AD), to be rated out of 5 grades (1, no problem; 2, slight problem; 3, some/moderate problem; 4, severe problem; 5, extreme problem).
Lumbar ROM from Baseline Lumbar ROM at each time point | Baseline (admission), 2 weeks after baseline, discharge (up to 14 weeks after baseline)
  Lumbar Range of Motion(ROM) (Flexion/Extension/Lateral flexion/Rotation) Pain upon movement in lumbar range of motion (ROM) will be assessed.
SLR from Baseline SLR at each time point | Baseline (admission), 2 weeks after baseline, discharge (up to 14 weeks after baseline)
  Straight Leg Raise test(SLR) The straight leg raise(SLR)is a test done during a physical examination to determine whether a patient with low back pain has an underlying herniated disc, often located at L5 (fifth lumbar spinal nerve).
  If the patient experiences sciatic pain when the straight leg is at an angle of between 30 and 70 degrees, then the test is positive and a herniated disk is a possible cause of the pain.[3] A negative test suggests a likely different cause for back pain.
AE | up to 14 weeks after baseline
  Adverse events(AE) Physicians will monitor and record any unexpected or unintended patient reaction to integrative korean medicine at each visit. Adverse events (AEs) associated with integrative korean medicine will include, but not be limited to, AEs anticipated from previous reports of korean medicine, and will stay open to all possibilities taking into consideration other potential, unknown AEs.
NRS change from Baseline NRS at each timepoint | Baseline (admission), 2 weeks after baseline, 6 months after baseline
  Numeric rating scale (NRS) of low back pain, and radiating leg pain In pain measurement using NRS, patients are asked to rate their pain by selecting a number from 0 to 10 that best represents their pain severity between the anchors of 0 which indicates 'no pain', and 10 which indicates 'worst pain possible'.
ODI change from Baseline ODI at each timepoint | Baseline (admission), 2 weeks after baseline, 6 months after baseline
  Oswestry Disability Index(ODI) The ODI evaluates functional impairment and is a 10-item questionnaire developed to assess the level of disability due to back pain. Each item is graded into 6 levels, each representing a score of 0-5. Higher scores indicate greater limitation relating to back pain.

CONTACTS AND LOCATIONS:
Overall Officials: HYUN WOO CHO, PhD, Principal Investigator — Haeundae Jaseng Hospital of Korean Medicine
Locations (4):
- South Korea (4):
  - Bucheon Jaseng Hospital of Korean Medicine, Bucheon-si, Gyeonggi Province
  - Haeundae Jaseng Hospital of Korean Medicine, Busan
  - Daejeon Jaseng Hospital of Korean Medicine, Daejeon
  - Jaseng Hospital of Korean Medicine, Seoul

IPD SHARING:
Plan to Share IPD: Undecided